CLINICAL TRIAL: NCT01313780
Title: A 4-week Multicentre, Randomized, Open Label, Parallel Group, Active Control Phase IV Study to Evaluate Efficacy and Safety of Oxycodone/Naloxone in Comparison With Oxycontin in Korean Patients With Cancer Pain(TOP)
Brief Title: A Study to Evaluate Efficacy and Safety of Oxycodone/Naloxone Compared to OxyContin in Korean Cancer Patients
Acronym: TOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXN10-KR-002
Record Dates: First submitted 2011-03-08; First posted 2011-03-14 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: cancer related pain
MeSH Terms: conditions — Neoplasms; Cancer Pain | interventions — Oxycodone; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 'Oxycodone/Naloxone' (Experimental): Trade name is Targin(fixed combination drug).
  Interventions: Drug: Oxycodone/Naloxone
- Oxycodone (Active Comparator): Trade name is Oxycontin(single compound).
  Interventions: Drug: Oxycodone(single compound)

INTERVENTIONS:
Drug: Oxycodone/Naloxone — Dose and administration : Upto 40mg B.I.D per daily.
  Other Names: Targin(fixed combination drug)
  Arms: 'Oxycodone/Naloxone'
Drug: Oxycodone(single compound) — Dose and administration : Upto 40mg B.I.D per daily.
  Other Names: Oxycontin
  Arms: Oxycodone

SUMMARY:
Objectives:

To prove non-inferiority of Targin compared to Oxycontin in terms of change of pain intensity

1. Primary objective: Change of pain intensity (NRS 0-10) score (average pain over 24 hours obtained each evening) within 4 weeks
2. Secondary objectives: Bowel Habit (worsening/no change/improving), Total dose and frequency of rescue medication, Quality of Life (QOL; EORTC QLQ-C30), Duration to need of laxative use and Adverse events

DETAILED DESCRIPTION:
This will be a 4-week multicentre, randomized, open label, parallel group, active control study to evaluate efficacy and safety of Targin in comparison with Oxycontin in Korean patients with cancer pain who are administered weak opioid or naïve patients including patient not on the long term strong opioid medication within 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female cancer patients 20 years of age or older
2. Cancer related pain that requires treatment with continuous around-the-clock strong opioid analgesic
3. Moderate to severe pain intensity(NRS pain score 4)
4. Opioid naïve patients or patients not treated with strong opioids(except PRN) within 4 weeks or patients who has been on weak opioids
5. Subject who provide signed and dated written voluntary informed consent

Exclusion Criteria:

1. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant. UNLESS they are:

   * women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner
   * women shoes partners have been sterilized by vasectomy or other means
   * two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
2. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test.
3. Have previously received treatment with Targin or Oxycontin within 4weeks(28days) of screening periods(including PRN)
4. If subjects started first cycle of chemotherapy during the 2 weeks before the screening visit or during the study, they should be excluded from the study.

   And If the chemotherapy regimen or dosage to be planned to change during the study, the subjects should be excluded from the study.
5. Patient who is administered laxatives with stable dose for more than 1 week
6. Patient with evidence of significant structural/functional abnormalities of GI tract which is not appropriate for oral medicine administration. Any history of hypersensitivity to Oxycodone and Naloxone
7. Patients with significant respiratory depression
8. Patients with acute or severe bronchial asthma or hypercarbia
9. Any patient who has or is suspected of having paralytic ileus
10. Severe Chronic obstructive pulmonary disease, pulmonary heart disease
11. Targin product contains lactose. Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption should not take
12. Patients with moderate and severe hepatic impairment
13. Abnormal aspartate aminotransferase (AST; SGOT), alanine aminotransferase (ALT; SGPT), or alkaline phosphatase levels (>2.5 times the upper limit of normal, it is allowed >5 times the upper limit of normal in case of transition in liver) or an abnormal total bilirubin and/or creatinine level(s) (greater than 1.5 times the upper limit of normal)
14. Any situation where opioids are contraindicated
15. Major surgery within 1 month prior to screening or planned surgery
16. Mainly pain originated other than cancer or cancer related conditions (eg. Musculoskeletal pain, inflammatory pain, diabetic polyneuropathy)
17. Patients with known or suspected unstable brain metastases or spinal cord compression that may require changes in steroid treatment throughout the duration of the study
18. Patients with uncontrolled seizures
19. Requiring interventional treatment for pain such as neurodestructive procedure or regional infusion
20. With a history of alcohol abuse within 6 months of screening
21. With a history of illicit drug abuse within 6 months of screening
22. Patients with increased intracranial pressure
23. In the investigator's opinion, subjects who are receiving hypnotics or other central nervous system (CNS) depressants that may pose a risk of additional CNS depression with opioid study medication
24. Patients with myxoedema, not adequately treated hypothyroidism or Addison's disease
25. Patients receiving opioid substitution therapy for opioid addiction (e.g. methadone or buprenorphine)
26. Patients with evidence of clinically significant gastrointestinal disease (e.g. paralytic ileus, peritoneal carcinosis), significant structural abnormalities of the gastrointestinal tract (e.g. scarring, obstruction etc) either related or not related to the underlying cancer or disease progression
27. Patients suffering from diarrhea and/or opioid withdrawal
28. With a disability that may prevent the patient from completing all study requirements and in particular, interfere with 24hrs pain intensity score
29. Clinically significant impairment of cardiovascular, respiratory and renal function
30. Patient who needs acute dose titration or whose pain intensity fluctuate significantly in a short period according to investigator's judgment
31. Having used other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim, M.D, Principal Investigator — Asan Medical Center; Ahn, M.D, Principal Investigator — Samsung Medical Center; Kim, M.D, Principal Investigator — National Cancer Center; Kim, M.D, Principal Investigator — SMG-SNU Boramae Medical Center; Lee, M.D, Principal Investigator — Shinchone Yonsei Severance Medical Center; Kang Jugnhoon, Principal Investigator — Kyungsang University Hospital; Lee Kyunghee, MD, Principal Investigator — Youngnam Univ. Hospital; Yoon Hwanjung, MD, Principal Investigator — Chungnam University Hospital
Locations (1):
- AMC, Seoul, Pungnap-dong, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee KH, Kim TW, Kang JH, Kim JS, Ahn JS, Kim SY, Yun HJ, Eum YJ, Koh SA, Kim MK, Hong YS, Kim JE, Lee GW. Efficacy and safety of controlled-release oxycodone/naloxone versus controlled-release oxycodone in Korean patients with cancer-related pain: a randomized controlled trial. Chin J Cancer. 2017 Sep 11;36(1):74. doi: 10.1186/s40880-017-0241-4. PMID 28893309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ITT set(Safety analysis) was 128(64:64) patients, but Missing primary efficacy data: 7 patients, Violation of inclusion/exclusion criteria: 4. So, FAS(Efficacy analysis) set population was 117(oxycodone/naloxone group: 58: Oxycodone: 59).
Groups:
- Oxycodone and Naloxone: Trade name is TARGIN. Daily dose can be titrated up to 40mg B.I.D.
- Oxycodone: Trade name is Oxycontin. Daily dose can be titrated up to 40mg B.I.D.
Period: Overall Study
Arm/Group | Oxycodone and Naloxone | Oxycodone
Started | 58 (FAS) | 59 (FAS)
Completed | 33 (PPS) | 31 (PPS)
Not Completed | 25 | 28
Not completed — Lack of Efficacy | 4 | 2
Not completed — Adverse Event | 6 | 11
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Protocol Violation | 10 | 4
Not completed — missing data | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone and Naloxone | Oxycodone | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Customized [Number; unit: participants]
  <39years | 1 | 3 | 4
  40~49years | 7 | 5 | 12
  50~59years | 19 | 17 | 36
  60~69 years | 14 | 23 | 37
  70~79 years | 17 | 11 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 43 | 39 | 82
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 58 | 59 | 117

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain Intensity From Baseline(visit1) to 4weeks.(visit3)
Description: Change of pain intensity from 0(No pain) to 10(worst pain imaginable) after 4 weeks treatment .
Time Frame: 4weeks
Population: Analysis of FAS: 117.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone and Naloxone | Oxycodone
Number analyzed (Participants) | 58 | 59
units on a scale | 1.586 (2.217) | 1.559 (2.215)

2. Secondary Outcome: Change in Bowel Habits.
Description: The change of bowel habits from baseline (Visit 1) in bowel habits at Week 4 was investigated, and was categorized as 'improved', 'unchanged', and 'worsened'.
Time Frame: 4 weeks
Population: FAS analysis, but Oxycodone/naloxone group was missed 15 patients data and Oxycodone group was missed 23 patients data.
Measure: Number; unit: participants
Arm/Group | Oxycodone and Naloxone | Oxycodone
Number analyzed (Participants) | 43 | 36
participants
  Unchanged | 31 | 20
  worsened | 7 | 11
  Improved | 5 | 5

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Subjects will be asked to voluntarily report adverse event information any time, and the information will be also checked at phone visits and regular visits during the treatment period through interviews and medical examination by the investigator.
Groups:
- Oxycodone and Naloxone: Oxycodone and naloxone: Trade name is TARGIN.
- Oxycodone: oxycodone : Trade name is Oxycontin
Arm/Group | Oxycodone and Naloxone | Oxycodone
Serious Adverse Events (participants affected / at risk) | 15/64 | 28/64
Other Adverse Events (participants affected / at risk) | 55/64 | 57/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone and Naloxone (N=64) | Oxycodone (N=64)
anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
leukocytosis (Investigations) | 0 (0) | 1 (1)
neutropenia (Investigations) | 1 (1) | 0 (0)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
General condition worse (General disorders) | 0 (0) | 1 (1)
Sweating (General disorders) | 0 (0) | 1 (1)
Disorder of adrenal gland (Endocrine disorders) | 0 (0) | 1 (1)
aggravated abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1)
ascitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
protruding mass in oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
rectal cancer progression (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
worsening vomitting (Gastrointestinal disorders) | 0 (0) | 1 (2)
cancer progression(gallbladder) (Hepatobiliary disorders) | 1 (1) | 0 (0)
jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
progress of disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 2 (2) | 0 (0)
left neck neoplasm (lymph node) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
leg edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Elevation of ALT (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Elevation of AST (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Electro imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
lower extremity weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Rt. Clavicle metasis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anxiety (Nervous system disorders) | 0 (0) | 1 (1)
both, limb numbness (Nervous system disorders) | 0 (0) | 1 (2)
delirium (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
hand tremor (Nervous system disorders) | 0 (0) | 1 (1)
HYPERALGESIA (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (2)
somnolence (Nervous system disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2)
Pain aggresive (General disorders) | 0 (0) | 1 (1)
stent insertion site pain (Surgical and medical procedures) | 0 (0) | 1 (1)
aggravation of lung metastasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cancer proression(lung) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
obstruction, ureter (Renal and urinary disorders) | 1 (1) | 0 (0)
PCN malfunction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone and Naloxone (N=64) | Oxycodone (N=64)
anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Megablastic anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
cold sweating (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3) | 3 (3)
Fever (General disorders) | 1 (1) | 1 (1)
General condition worse (General disorders) | 0 (0) | 1 (1)
General weakness (General disorders) | 1 (2) | 0 (0)
Insomnia (Nervous system disorders) | 3 (3) | 1 (1)
night fever (General disorders) | 1 (1) | 0 (0)
Sweating (General disorders) | 0 (0) | 1 (1)
Sweating (diaphoresis) (General disorders) | 0 (0) | 1 (1)
Weight loss (General disorders) | 1 (2) | 0 (0)
itching sense(WB) (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (5)
skin lesion on ear (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
skin nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
whole body itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Disorder of adrenal gland (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal palpable mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
aggravated abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 8 (14) | 4 (4)
ascitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 30 (36) | 35 (37)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 1 (1)
heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (11) | 18 (19)
protruding mass in oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
rectal cancer progression (Gastrointestinal disorders) | 0 (0) | 1 (1)
reducing oral intake (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (9) | 7 (7)
worsening vomitting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hematochezia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
hemoptysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
cancer progression(gallbladder) (Renal and urinary disorders) | 1 (1) | 0 (0)
jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
progress of disease (Hepatobiliary disorders) | 1 (1) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Edema ; both leg (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Edema of legs (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
left neck neoplasm (lymph node) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
leg edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 0 (0) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 0 (0) | 1 (1)
Calcium, serum-high (hypercalcemia) (Investigations) | 1 (1) | 0 (0)
Elevated creatininte (Investigations) | 1 (4) | 0 (0)
Elevation of ALT (Investigations) | 1 (1) | 0 (0)
Elevation of AST (Investigations) | 1 (1) | 0 (0)
Glucose, serum-high (hyperglycemia) (Investigations) | 1 (1) | 0 (0)
Glucose, serum-low (hypoglycemia) (Investigations) | 2 (5) | 0 (0)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Liver enzyme increase (Investigations) | 1 (1) | 0 (0)
Potassium, serum-high (hyperkalemia) (Investigations) | 1 (3) | 1 (1)
Potassium, serum-low (hypokalemia) (Investigations) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Investigations) | 1 (1) | 0 (0)
Electro imbalance (Investigations) | 0 (0) | 1 (2)
lower extremity weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
progress of disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rt. Clavicle metasis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 2 (2)
both, limb numbness (Nervous system disorders) | 0 (0) | 1 (2)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
delirium (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 6 (7) | 14 (15)
hand tremor (Nervous system disorders) | 0 (0) | 1 (1)
head trauma (Nervous system disorders) | 1 (1) | 0 (0)
HYPERALGESIA (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0)
peripheral neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (2)
somnolence (Nervous system disorders) | 3 (3) | 3 (3)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dysuria (Renal and urinary disorders) | 3 (3) | 3 (3)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
headache (Nervous system disorders) | 1 (1) | 2 (2)
low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
lt shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
lt.knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain (Right Upper Quadrant) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain ; abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain aggresive (General disorders) | 0 (0) | 1 (1)
pantalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
peivic pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
stent insertion site pain (Surgical and medical procedures) | 0 (0) | 1 (1)
worsing abdomen pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
aggravation of lung metastasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cancer proression(lung) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Dyspnea on exercise (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
progress of disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Difficult urination (Renal and urinary disorders) | 0 (0) | 1 (1)
obstruction, ureter (Renal and urinary disorders) | 1 (1) | 0 (0)
PCN malfunction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Voiding difficulty (Renal and urinary disorders) | 1 (1) | 0 (0)
Infusion related reaction (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No